CLINICAL TRIAL: NCT04904991
Title: Three-month Chan-Chung Qigong Program in Improving Physical Functional Performance and Quality of Life in Cognitive Impairment Patients
Brief Title: Three-month Chan-Chung Qigong Improves Physical Function Performance and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Hsu Chin-yun, Head Nurse, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-105-05-133
Record Dates: First submitted 2020-12-13; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Cognitive Dysfunction; Cognitive Aging; Grip; Exercise Training; Physical Endurance; Cognitive Decline
Keywords: Cognitive inpairment; Qigong / Exercise; Muscle strength /endurance; Quality of life; Physical activity
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study randomized controlled trial with four repeated measurements was conducted between Apply 2016 and October 2017. Participants in the Qigong group were given a structured program about Chan-Chung qigong for 3 months; those in the control group received usual care for cognitive impairment during the same study period. The intervention effects were measured by muscular strength, muscular endurance, and 6-min walk distance at baseline, Month 1, Month 2, and Month 3. In addition, QoL was measured at baseline and Month 3.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qigong group (Experimental): Participants in the Qigong group were given a structured program about Chan-Chung qigong for 3 months which was a modified form of the manual of Chan-Chuang qigong (Yeh et al., 2006), to tailor to patients with cognitive impairment. The Chan-Chuang qigong program included warmup prior to qigong practice, preparation for qigong practice . The movements should be repeated and maintained for 10 minutes per time, 3 time a day .
  Interventions: Procedure: Chan-Chuang qigong
- Control group (No Intervention): those in the control group received usual care for cognitive impairment during the same study period.

INTERVENTIONS:
Procedure: Chan-Chuang qigong — This study applied the Chan-Chuang qigong program, which was a modified form of the manual of Chan-Chuang qigong (Yeh et al., 2006), to tailor to patients with cognitive impairment. The Chan-Chuang qigong program included warmup prior to qigong practice, preparation for qigong practice, core qigong of four moves, and cool down after qigong practice.
  The movements should be repeated and maintained for 10 minutes per time, 3 time a day (Yeh et al., 2006), totally 90 minutes per week, for 3 months. The guideline booklet of Chan-Chuang qigong (Chen et al., 2019; Chuang, Yeh, & Chung, 2017) was modified and provided to the participants, which had major sections of introduction to qigong, preparation and precautions, practical procedures with description and photos, normal physical reactions from practicing core Chan-Chuang qigong, precautions of daily life, a confirmation sheet, and a checklist of qigong performance.
  Other Names: qigong group
  Arms: Qigong group

SUMMARY:
The purpose of this study aimed to evaluate the effect of the three-month Chan-Chung qigong program in improving physical functional performance and quality of life in patients with mild to moderate cognitive impairments.A quasi-experimental design was adopted. Subjects were recruited from cognitive impairments outpatients these subjects,41were assigned to the control group and 41 to the experimental group in which Chan-Chuang qigong was administered.

DETAILED DESCRIPTION:
This study randomized controlled trial with four repeated measurements was conducted between Apply 2016 and October 2017. Participants in the Qigong group were given a structured program about Chan-Chung qigong for 3 months; those in the control group received usual care for cognitive impairment during the same study period. The intervention effects were measured by muscular strength, muscular endurance, and 6-min walk distance at baseline, Month 1, Month 2, and Month 3. In addition, QoL was measured at baseline and Month 3.

ELIGIBILITY:
Inclusion Criteria:

* Participants invited in this study were aged more than 60 years, diagnosed with the Clinical Dementia Rating (CDR) ≦1, able to communicate, free to stand and walk, and willing to participate this study.

Exclusion Criteria:

* The exclusion criteria were as followings: use of hormone drugs, brain trauma, head surgery, vitamin B12 deficiency, decreased memory and judgment due to hypothyroidism or malnutrition with medical contraindications for exercise, and practicing qigong or exercise regularly.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2017-11-04 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
The findings of this study indicate Chan-Chuang qigong improved physical function performance with cognitive impairment. | 3 months
  this study considered the influences of cognition status and changes. After the intervention measures were implemented, the Qigong group had significant differences in physiological function, muscle endurance, and cardiopulmonary fitness compared with the control group.
There was no significant between-group difference in the physical and mental components at baseline. | 3 months
  However, a significant between-group difference was in the physical , not mental, component on Month 3. In addition, no significant within-group difference in either Qigong or control group